CLINICAL TRIAL: NCT04616755
Title: Stability of Maxillary Anterior Teeth After Two Years of Retention in Adolescents - A Randomized Controlled Trial Comparing Two Bonded and a Vacuum-formed Retainer
Brief Title: Stability of Maxillary Anterior Teeth After Two Years of Retention in Adolescents Comparing Two Bonded and a Vacuum-formed Retainer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kronoberg County Council (Other Government)
Collaborators: Malmö University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Region Kronoberg
Record Dates: First submitted 2020-10-23; First posted 2020-11-05 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Orthodontic Appliance Complication
Keywords: Retention devices; Relapse; Maxillary incisors; Irregularity
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Intervention Model Description: Three groups with different retention devices
Who Masked: Outcomes Assessor
Masking Description: All study casts will be scanned without name just with a number and assessor do not know which group they belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bonded retainer 13-23 (Active Comparator): This group have bonded retainer behind six front teeth in the maxilla to keep front teeth stable.
  Interventions: Other: Measuring changes of Little´s irregularity index ( sum of 5 contact point discrepancies together) measured in mm 2 years after retention have been I place.
- Bonded retainer 12-22 (Active Comparator): This group have bonded retainer behind four front teeth in the maxilla to keep front teeth stable.
  Interventions: Other: Measuring changes of Little´s irregularity index ( sum of 5 contact point discrepancies together) measured in mm 2 years after retention have been I place.
- Vacuum-formed retainer (Active Comparator): This group have Vacuum-formed retainer covering all erupted teeth in maxilla to keep front teeth stable
  Interventions: Other: Measuring changes of Little´s irregularity index ( sum of 5 contact point discrepancies together) measured in mm 2 years after retention have been I place.

INTERVENTIONS:
Other: Measuring changes of Little´s irregularity index ( sum of 5 contact point discrepancies together) measured in mm 2 years after retention have been I place. — Measuring changes occurred under 2 years which the retention devices have been in place between the groups
  Other Names: Measuring changes of 5 single Contact point displacements in mm 2 years after retention have been I place.

SUMMARY:
After orthodontic treatment 3 different retention devices will be compared.Thirty patients in each group; Group 1) Bonded retainer 13-23, Group 2)Bonded retainer 12-22 and Group 3) Vacuum-formed retainer covering all erupted teeth in the maxilla. Retention capacity between these three devices will be compared after 2 years of retention by measuring Contact Point displacements (CPD) between 6 anterior teeth and sum of 5 anterior CPDs called Little´s Irregularity Index (LII).

DETAILED DESCRIPTION:
Studies have shown that esthetics, no doubt, is the major motivating factor for orthodontic treatment both in adults and adolescents.Orthodontic relapses are usually described as changes toward the pretreatment status. These changes occur very fast if the teeth are not kept in their new position. That is the reason why, after orthodontic treatment, the result must be stabilized by some kind of retention device to prevent relapse. However, after this first period of remodeling of periodontal structures, comes the later period of changes.

Relapse in aesthetic zone (Anterior teeth), is the major reason why patients are dissatisfied with the results and seek for retreatment. There is a gap in our knowledge which kind of retention device is more effective to stabilize achieved alignment after orthodontic treatment.

This randomized clinical trial, tries to answer to that question. The investigators shall compare three different retention devices and measure changes after 2 years when retention devices have been in place and later compare the long-term results when the retainers have been removed after 2 years of retention (future study 5 years ptstretention).

Randomization Three months before the estimated removal of the fixed appliances, the patients will be invited to take part in the trial. After gaining informed consent from the patient and their custodians, the patients are randomly allocated to one of the three retention groups as follow: A) bonded retainer 13-23, B) bonded retainer 12-22 and C) removable vacuum-formed retainer (VFR) covering the maxillary teeth including the second molars. The randomization process is prepared by an independent person and carried out by three staff members not involved in the trial. The randomization uses blocks of 30. The randomization notes is delivered in a sealed opaque envelope each. Every new participant picked an envelope and reveal the group assignment by opening the envelope. Recruitment is ongoing until the total number of participants meet the estimated sample size.

ELIGIBILITY:
Inclusion Criteria:

* Young children age between 11 to 19 years old undergone orthodontic treatment.

Exclusion Criteria:

* Syndrome patients
* Skeletal discrepancy
* missing maxillary anterior teeth
* Adults

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Changes in LII (sum of 5 contact point discrepancy)among 6 maxillary front teeth | 2 years after retention device in place
  Sum of five single contact points of maxillary anterior teeth
Changes in CPD | 2 years after retention device in place
  Changes in single contact point discrepancy of five maxillary anterior teeth

SECONDARY OUTCOMES:
Intercanine distance | 2 years after retention device in place
  Measuring the distance between top of the canines in maxilla
Intermolar distance | 2 years after retention device in place
  Measuring the distance between cusp tips of first molars

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naraghi S, Ganzer N, Bondemark L, Sonesson M. Stability of maxillary anterior teeth during retention and 1 year after removal of retention-an RCT on adolescents retained with two different bonded retainers and a vacuum-formed retainer. Eur J Orthod. 2023 Nov 30;45(6):629-636. doi: 10.1093/ejo/cjad020. PMID 37119264
- [Derived] Sonesson M, Naraghi S, Bondemark L. Cost analysis of two types of fixed maxillary retainers and a removable vacuum-formed maxillary retainer: a randomized controlled trial. Eur J Orthod. 2022 Mar 30;44(2):197-202. doi: 10.1093/ejo/cjab080. PMID 35021204
- [Derived] Naraghi S, Ganzer N, Bondemark L, Sonesson M. Stability of maxillary anterior teeth after 2 years of retention in adolescents: a randomized controlled trial comparing two bonded and a vacuum-formed retainer. Eur J Orthod. 2021 Apr 3;43(2):152-158. doi: 10.1093/ejo/cjaa077. PMID 33351886